CLINICAL TRIAL: NCT03575910
Title: HEARTBiT: A Novel Multi-Marker Blood Test for Management of Acute Cardiac Allograft Rejection
Brief Title: HEARTBiT: Multi-Marker Blood Test for Acute Cardiac Transplant Rejection
Acronym: HEARTBiT
Status: Active, not recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); PROOF Centre of Excellence (Unknown); Duke University (Other); University of Nebraska (Other); Toronto General Hospital (Other); St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Scott Tebbutt, Professor, University of British Columbia
Other Study IDs: PROOF
Record Dates: First submitted 2018-06-19; First posted 2018-07-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Heart Transplant Failure and Rejection; Heart Failure; Heart Diseases; Heart Failure，Congestive; Transplant; Failure, Heart; Transplant Failure
Keywords: Heart; Transplantation; Acute cardiac rejection; Biomarkers; Genomics
MeSH Terms: conditions — Rejection, Psychology; Heart Failure; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples to be collected in four (4) tubes (approx. 15mL or 3 teaspoons) consisting of:
  1. 1 - 6 mL lavender top (EDTA) tube (plasma)
  2. 1 - 4 mL red top tube (serum)
  3. 2 - 2.5 mL PAXgene tubes (RNA)
  Blood processing (fractionation) of plasma and serum tubes following SOP guidelines will result in collection of:
  8 - 0.5mL plasma aliquots
  1 - 0.5mL buffy coat DNA sample 6 - 0.5mL serum aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Acute Rejection (AR): Heart transplant patients diagnosed with an ISHLT grade 2R or 3R via endomyocardial biopsy.
- Mild Rejection (MR): Heart transplant patients diagnosed with an ISHLT grade 1R via endomyocardial biopsy.
- Non-Rejection (NR): Heart transplant patients diagnosed with an ISHLT grade 0R via endomyocardial biopsy.

SUMMARY:
Heart transplantation is a life saving therapy for people with end stage heart failure. Acute rejection, a process where the immune system recognizes the transplanted heart as foreign and mounts a response against it, remains a clinical problem despite improvements in immunosuppressive drugs. Acute rejection occurs in 20-30% of patients within the first 3 months post-transplant, and is currently detected by highly invasive heart tissue biopsies that happen 12-15 times in the first year post-transplant. Replacing the biopsy with a simple blood test is of utmost value to patients and will reduce healthcare costs. The goal of our project is to develop a new blood test to monitor heart transplant rejection. Advances in biotechnology have enabled simultaneous measurement of many molecules (e.g., proteins, nucleic acids) in blood, driving the development of new diagnostics. Our team is a leader in using computational tools to combine information from numerous biological molecules and clinical data to generate "biomarker panels" that are more powerful than existing diagnostic tests. Our sophisticated analytic methods has recently derived HEARTBiT, a promising test of acute rejection comprising 9 RNA biomarkers, from the measurement of 30,000 blood molecules in 150 Canadian heart transplant patients. Our objective is to study a custom-built HEARTBiT test in a setting and on a technology that enable clinical adoption. We will evaluate the new test on 400 new patients from 5 North American transplant centres. We will also track patients' HEARTBiT scores over time to help predict future rejection, and explore use of proteins and micoRNAs to improve HEARTBiT. Our work will provide the basis for a future clinical trial. The significance of this work rests in that it will provide a tool to identify acute cardiac rejection in a fast, accurate, cost-effective and minimally invasive manner, allowing for facile long-term monitoring and therapy tailoring for heart transplant patients.

DETAILED DESCRIPTION:
Rationale:

Cardiac transplantation remains the main intervention for those with end-stage heart failure. Maintenance immunosuppression is given to all transplant recipients to prevent acute rejection and loss of the allograft. Despite great improvements in immunosuppressive therapies, acute rejection remains a clinical problem and occurs at varying severity in 20-30% of patients within the first 3 months post-transplant. Timely detection of moderate rejection allows for treatment to be modified, preventing organ damage, graft failure and patient death. The current method to monitor for rejection remains the endomyocardial biopsy (EMB), a highly invasive and costly procedure that poses physical risks and emotional stress to patients, who must undergo 12-15 such tests during the first year post-transplant. EMB detects rejection only when tissue damage has occurred, and lacks sensitivity as it provides information about tiny pieces of the endomyocardium. Clearly, patients and clinicians would benefit from an effective, cheaper, less invasive diagnostic test that can indicate when an EMB is not needed.

Our team used unbiased omics strategies and computational tools to identify potential biomarkers of treatable acute rejection (ISHLT grade 2R or higher) in peripheral blood. We hypothesize that there are distinctive RNA and protein signatures in blood that can be developed into a simple test to accurately indicate when heart transplant patients do not require EMB, and that studying these biomarkers in a clinically relevant setting will facilitate clinical adoption.

Our Specific Aims are to:

1. Evaluate the performance of HEARTBiT, a custom 9-mRNA biomarker test developed on the NanoString platform, in an environment suitable for clinical translation, on >4000 newly collected samples from 400 patients across North America
2. Examine the biomarker panel score and individual biomarkers serially across the first year post-transplant to identify predictive signatures of rejection and characterize underlying biology
3. Develop and assess 5 promising protein biomarker candidates on NanoString, test 7 candidate miRNAs, and evaluate combinatorial RNA-protein classifier performance metrics to improve HEARTBiT

Expertise: Our team at the Centre of Excellence for Prevention of Organ Failure has over 10 years experience in computational analysis of omics and clinical data to create biomarker tests that out-perform current gold standards. Our Biomarkers in Transplantation (BiT) study has been continuously funded by competitive grants, philanthropy and industry between 2004-2017 and has generated many publications related to heart and kidney transplant rejection. Via our collaborators, we will have access to a Canadian Blood Services facility for testing our biomarkers, and patient samples from 5 major transplant sites (St. Paul's/Vancouver, Toronto, Nebraska, Newark Beth Israel, Duke).

Outcomes: The HEARTBiT test will be ready for clinical utility studies. The test will have significant clinical and socioeconomic value by reducing EMBs for transplant patients and enabling the tailoring of therapy. Insights into the biology of immune rejection will also be enhanced.

ELIGIBILITY:
Heart Transplant Subjects:

Inclusion Criteria

* recipients who are ≥ 19 years of age
* willing and able to provide informed consent

Exclusion Criteria

* recipients under 19 years of age
* recipients who have received multiple, different solid organ transplants (i.e. a heart and a kidney)
* recipients who are HIV positive
* recipients of organs from donors who test positive for HIV

Normal Subjects:

Inclusion Criteria

* all individuals who are ≥ 19 years of age
* willing and able to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is anticipated that up to 400 heart transplant recipients will be enrolled as participants. Given the prevalence of treatable AR observed at the recruiting sites, 40-50 AR and 350 NR/MR are expected, excluding the time course (first year post-transplant) samples. Additionally, we plan on enrolling 30 normal control subjects. Comparisons will be made between AR, MR, and NR samples from independent patients.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the HEARTBiT Biomarker Panel Score (BPS) between acute rejection and non-rejection/mild-rejection samples on the NanoString platform. | Within 5 years
  The performance of HEARTBiT, a custom 9-RNA biomarker assay developed on the NanoString platform, will be evaluated in an environment suitable for clinical translation using a sample size of ~4000 newly collected samples from 400 HT patients. Performance will be assessed by applying an algorithm that combines the quantitative data of the 9 RNA into a single BPS. This score aggregates the influence of all RNAs and will be associated with an estimated probability that AR is occurring in the transplant recipient. The algorithm will establish a single cutoff thus producing a final binary test result (AR or NR/MR), or, if possible, two cutoffs to separate AR, MR and NR as ordered variables.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tebbutt, PhD, Principal Investigator — University of British Columbia
Locations (4):
- University of Nebraska Medical Center, Omaha, Nebraska, United States
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital UHN, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sukma Dewi I, Gidlof O, Hollander Z, Lam KK, Benson MD, Braun OO, Nilsson J, Tebbutt SJ, Ng RT, Ohman J, McManus BM, Smith JG. Immunological Serum Protein Profiles for Noninvasive Detection of Acute Cellular Rejection After Heart Transplantation. J Am Coll Cardiol. 2017 Dec 12;70(23):2946-2947. doi: 10.1016/j.jacc.2017.10.012. No abstract available. PMID 29216990
- [Background] Toma M, Mak GJ, Chen V, Hollander Z, Shannon CP, Lam KKY, Ng RT, Tebbutt SJ, Wilson-McManus JE, Ignaszewski A, Anderson T, Dyck JRB, Howlett J, Ezekowitz J, McManus BM, Oudit GY. Differentiating heart failure phenotypes using sex-specific transcriptomic and proteomic biomarker panels. ESC Heart Fail. 2017 Aug;4(3):301-311. doi: 10.1002/ehf2.12136. Epub 2017 Mar 4. PMID 28772032
- [Background] Sukma Dewi I, Hollander Z, Lam KK, McManus JW, Tebbutt SJ, Ng RT, Keown PA, McMaster RW, McManus BM, Gidlof O, Ohman J. Association of Serum MiR-142-3p and MiR-101-3p Levels with Acute Cellular Rejection after Heart Transplantation. PLoS One. 2017 Jan 26;12(1):e0170842. doi: 10.1371/journal.pone.0170842. eCollection 2017. PMID 28125729
- [Background] Sukma Dewi I, Celik S, Karlsson A, Hollander Z, Lam K, McManus JW, Tebbutt S, Ng R, Keown P, McMaster R, McManus B, Ohman J, Gidlof O. Exosomal miR-142-3p is increased during cardiac allograft rejection and augments vascular permeability through down-regulation of endothelial RAB11FIP2 expression. Cardiovasc Res. 2017 Apr 1;113(5):440-452. doi: 10.1093/cvr/cvw244. PMID 28073833
- [Background] Hollander Z, Lazarova M, Lam KK, Ignaszewski A, Oudit GY, Dyck JR, Schreiner G, Pauwels J, Chen V, Cohen Freue GV, Ng RT, Wilson-McManus JE, Balshaw R, Tebbutt SJ, McMaster RW, Keown PA, McManus BM; NCE CECR PROOF Prevention of Organ Failure (PROOF) Centre of Excellence. Proteomic biomarkers of recovered heart function. Eur J Heart Fail. 2014 May;16(5):551-9. doi: 10.1002/ejhf.65. Epub 2014 Feb 23. PMID 24574204
- [Background] Shin H, Gunther O, Hollander Z, Wilson-McManus JE, Ng RT, Balshaw R, Keown PA, McMaster R, McManus BM, Isbel NM, Knoll G, Tebbutt SJ. Longitudinal analysis of whole blood transcriptomes to explore molecular signatures associated with acute renal allograft rejection. Bioinform Biol Insights. 2014 Jan 22;8:17-33. doi: 10.4137/BBI.S13376.. eCollection 2014. PMID 24526836
- [Background] Cohen Freue GV, Meredith A, Smith D, Bergman A, Sasaki M, Lam KK, Hollander Z, Opushneva N, Takhar M, Lin D, Wilson-McManus J, Balshaw R, Keown PA, Borchers CH, McManus B, Ng RT, McMaster WR; Biomarkers in Transplantation and the NCE CECR Prevention of Organ Failure Centre of Excellence Teams. Computational biomarker pipeline from discovery to clinical implementation: plasma proteomic biomarkers for cardiac transplantation. PLoS Comput Biol. 2013 Apr;9(4):e1002963. doi: 10.1371/journal.pcbi.1002963. Epub 2013 Apr 4. PMID 23592955
- [Background] Hollander Z, Chen V, Sidhu K, Lin D, Ng RT, Balshaw R, Cohen-Freue GV, Ignaszewski A, Imai C, Kaan A, Tebbutt SJ, Wilson-McManus JE, McMaster RW, Keown PA, McManus BM; NCE CECR PROOF Centre of Excellence. Predicting acute cardiac rejection from donor heart and pre-transplant recipient blood gene expression. J Heart Lung Transplant. 2013 Feb;32(2):259-65. doi: 10.1016/j.healun.2012.11.008. Epub 2012 Dec 21. PMID 23265908
- [Background] Shannon CP, Hollander Z, Wilson-McManus J, Balshaw R, Ng RT, McMaster R, McManus BM, Keown PA, Tebbutt SJ. White blood cell differentials enrich whole blood expression data in the context of acute cardiac allograft rejection. Bioinform Biol Insights. 2012;6:49-61. doi: 10.4137/BBI.S9197. Epub 2012 Apr 10. PMID 22550401
- [Background] Lin D, Hollander Z, Meredith A, Stadnick E, Sasaki M, Cohen Freue G, Qasimi P, Mui A, Ng RT, Balshaw R, Wilson-McManus JE, Wishart D, Hau D, Keown PA, McMaster R, McManus BM; Biomarkers in Transplantation Team; NCE CECR PROOF Centre of Excellence. Molecular signatures of end-stage heart failure. J Card Fail. 2011 Oct;17(10):867-74. doi: 10.1016/j.cardfail.2011.07.001. Epub 2011 Sep 3. PMID 21962426
- [Background] Hollander Z, Lin D, Chen V, Ng R, Wilson-McManus J, Ignaszewski A, Cohen Freue G, Balshaw R, Mui A, McMaster R, Keown PA, McManus BM; NCE CECR PROOF Centre of Excellence. Whole blood biomarkers of acute cardiac allograft rejection: double-crossing the biopsy. Transplantation. 2010 Dec 27;90(12):1388-93. doi: 10.1097/TP.0b013e3182003df6. PMID 21076371
- [Background] Lin D, Hollander Z, Ng RT, Imai C, Ignaszewski A, Balshaw R, Freue GC, Wilson-McManus JE, Qasimi P, Meredith A, Mui A, Triche T, McMaster R, Keown PA, McManus BM; Biomarkers in Transplantation Team; NCE CECR Centre of Excellence for the Prevention of Organ Failure. Whole blood genomic biomarkers of acute cardiac allograft rejection. J Heart Lung Transplant. 2009 Sep;28(9):927-35. doi: 10.1016/j.healun.2009.04.025. PMID 19716046